CLINICAL TRIAL: NCT03139773
Title: Nutrition Intervention to Improve Energy Metabolism, Energy Intake, and Metabolic Response in Overweight and Obese School-aged Children
Brief Title: Nutrition Intervention to Measure Metabolic Response in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 15-09-094
Record Dates: First submitted 2017-03-08; First posted 2017-05-04 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Weight (Experimental): Received control breakfast beverage and breakfast beverage supplemented with omega-3 fatty acids.
  Interventions: Dietary Supplement: Control Breakfast Beverage; Dietary Supplement: Omega-3 Breakfast Beverage
- Overweight/Obese (Experimental): Received control breakfast beverage and breakfast beverage supplemented with omega-3 fatty acids.
  Interventions: Dietary Supplement: Control Breakfast Beverage; Dietary Supplement: Omega-3 Breakfast Beverage

INTERVENTIONS:
Dietary Supplement: Control Breakfast Beverage — Each participant consumes the breakfast beverage every morning before 10:00 am for 14 days.
Dietary Supplement: Omega-3 Breakfast Beverage — Each participant consumes the breakfast beverage every morning before 10:00 am for 14 days.

SUMMARY:
The long-term objective of this study is to determine if habitual consumption of high-quality protein at breakfast will lead to improved energy metabolism and decreased daily energy intake in normal weight and overweight children. The investigators hypothesize that increasing protein intake at breakfast will improve energy metabolism and reduce energy intake throughout the day in overweight/obese school-aged children. The significance of the study is that improving nutrient intake at breakfast can potentially lead to a future reduction in childhood obesity rates.

ELIGIBILITY:
Inclusion Criteria:

* Habitual breakfast consumer
* No known medical issues

Exclusion Criteria:

* Food allergies
* Medication
* Claustrophobic
* Dietary restrictions
* Picky eater (determined by parent/guardian)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
The effect of breakfast type on energy expenditure four hours postprandial | Change from baseline to four hours postprandial.
  Energy expenditure will be measured using indirect calorimetry via a TrueMax metabolic cart.
The effect of breakfast type on postprandial appetite | Change from baseline to four hours postprandial.
  Appetite assessment via visual analog scales
The effect of breakfast type on appetite hormone secretion | Change from baseline to four hours postprandial.
  Leptin, adiponectin, PYY, and CCK will be measured using ELISA method.
The effect of breakfast type on energy expenditure over 14 days of dietary adaptation. | Fourteen days
  Whole-body energy expenditure will be measured using doubly-labeled water method

SECONDARY OUTCOMES:
Metabolic health measures | Baseline and day 14 of each intervention
  Plasma insulin, glucose, lipids
Gut microbiota | Baseline and day 14 of each intervention
  Assessment of gut microbiome
Proteomic analysis using TMT labeling | Fasting levels at baseline
  Proteomic analysis of baseline samples

CONTACTS AND LOCATIONS:
Overall Officials: Jamie I Baum, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No